CLINICAL TRIAL: NCT05152186
Title: Comparison Between the Effect of Topical Tranexamic Acid Versus Hydrogen Peroxide on Perioperative Blood Loss in Elective Spine Surgeries
Brief Title: Compare Between the Effect of Topical Tranexamic Acid Versus Hydrogen Peroxide on Blood Loss in Spine Surgeries
Acronym: Bloodloss
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Nehal Kamal Mohamed, Assistant lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: blood loss in spine surgery
Record Dates: First submitted 2021-11-12; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Blood Loss
Keywords: Blood loss
MeSH Terms: conditions — Hemorrhage | interventions — Solutions; Therapeutic Irrigation; Disinfectants; Crystalloid Solutions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tranexamic acid (Active Comparator): Topical hemostatics as tranexamic acid or hydrogen peroxide in wound before skin closure to decrease perioperative blood loss
  Interventions: Drug: Topical Solution; Drug: Topical Foam; Other: Topical
- Hydrogen peroxide (Active Comparator): Topical hemostatics as hydrogen peroxide in wound before skin closure to decrease perioperative blood loss
  Interventions: Drug: Topical Solution; Drug: Topical Foam; Other: Topical
- Normal saline (Placebo Comparator): Hemostasis in spine surgery
  Interventions: Drug: Topical Solution; Drug: Topical Foam; Other: Topical

INTERVENTIONS:
Drug: Topical Solution — Topical administration
  Other Names: Irrigation
Drug: Topical Foam — Topical administration
  Other Names: Disinfectant
Other: Topical — Topical administration
  Other Names: Crystalloid

SUMMARY:
To evaluate the effectiveness of topical TXA in reducing blood loss compared to H2O2 wash.

The primary outcomes :

1. Estimation of Intraoperative blood loss and blood transfusion.
2. Recording Postoperative blood drainage.
3. Comparing Hemoglobin levels (pre and postoperative).

The secondary outcomes :

1. Surgical site infection (SSI)
2. Length of hospital stay.

DETAILED DESCRIPTION:
Spinal surgery is one of the most commonly performed neuro-surgeries worldwide. Massive blood loss occurs frequently and remains a challenge in complex spinal surgery. Significant intra and postoperative hemorrhage negatively affects patient outcomes by increasing coagulopathy, postoperative hematoma and anemia .The need for allogenic blood transfusions can lead to potential transfusion reactions and infections, in addition to increasing long-term mortality rates. There is an economic disadvantage associated with iatrogenic major blood loss relating to the direct costs of the blood products and intraoperative blood salvage technology and indirect costs of prolonged patient hospitalization and complication management .

Many efforts have focused on achieving better perioperative blood conservation, in particular through prophylactic intravenous administration of antifibrinolytic agents before and during major surgery. Intravenous administration of the inexpensive but highly effective drug as tranexamic acid (TXA) reduces perioperative hemorrhage and the need for blood transfusions by one third in major surgery, including spinal surgery, Included on the list of the World Health Organization (WHO) List of Essential Medicines, TXA has taken its place as a widely used hemostatic agent in the clinical setting .

Tranexamic acid is a synthetic analog of the amino acid lysine. It serves as an antifibrinolytic by reversibly binding four to five lysine receptor sites on plasminogen. This reduces conversion of plasminogen to plasmin, preventing fibrin degradation and preserving the framework of fibrin's matrix structure .Tranexamic acid has roughly eight times the antifibrinolytic activity of an older analogue, ε-aminocaproic acid. Tranexamic acid also directly inhibits the activity of plasmin with weak potency .

Hydrogen peroxide (H2O2) is an inexpensive and readily available option whose hemostatic and antiseptic properties have been separately confirmedin several previous studies .

ELIGIBILITY:
Inclusion Criteria:

* ASA: class II or III
* Sex: male and female
* Age: from 20 to 70 years.
* Type of operation: patient will undergo spinal surgery with a diagnosis of in place spinal trauma, thoracic or lumbar degenerative disease, such as spinal canal stenosis, disc herniation, spondylolisthesis, and/or degenerative scoliosis under general anesthesia.

Exclusion Criteria:

* Patients with history of thromboembolic disease or coagulopathy or hereditary bleeding disorders such as factor VIII deficiency, factor IX deficiency, and Von-Willebrand disease.
* Patients who were taking anticoagulants or antiplatelet drugs.
* Allergy or hypersensitivity to TXA.
* A dural tear accompanied by cerebrospinal fluid leakage detected intraoperatively.
* Spinal cord tumors, head trauma and penetrating spinal cord trauma.
* The use of intravenous TXA during the perioperative period .
* Infection at the operative site e.g T.B.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Blood loss estimation [NCT ID not yet assigned] | Within 48 hours
  Estimation of perioperative blood loss and need of blood transfusion, lab investigations pre and postoperative (hemoglobin (gm/dL), hematocrit (%), Prothrombin concentration (%), INR, platelets).
  * Recording Postoperative blood drainage (in ml). and Comparing Hemoglobin levels (pre and postoperative).

SECONDARY OUTCOMES:
Complications | 7 days
  Anaemia secondary to blood loss, surgical site infection , length of hospital stay (in days), complications of drugs used in procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Amani Khairy, Professor, Study Chair — Faculty of Medicine, Minia University; Sarah Mohamed, Lecturer, Study Director — Faculty of Medicine, Minia University; Walid Zidan, Lecturer, Study Director — Faculty of Medicine, Minia University; Nehal Kamal, Master, Principal Investigator — Faulty of medicine, Minia University
Locations (1):
- Minia University hospital, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qureshi R, Puvanesarajah V, Jain A, Hassanzadeh H. Perioperative Management of Blood Loss in Spine Surgery. Clin Spine Surg. 2017 Nov;30(9):383-388. doi: 10.1097/BSD.0000000000000532. PMID 28338491
- [Background] Hui S, Peng Y, Tao L, Wang S, Yang Y, Du Y, Zhang J, Zhuang Q; TARGETS study group. Tranexamic acid given into wound reduces postoperative drainage, blood loss, and hospital stay in spinal surgeries: a meta-analysis. J Orthop Surg Res. 2021 Jun 22;16(1):401. doi: 10.1186/s13018-021-02548-6. PMID 34158096